CLINICAL TRIAL: NCT06653634
Title: Optimizing Treatment for Children and Adolescents With Juvenile Idiopathic Arthritis in Sustained Remission: a Comparison of Three Treatment Strategies. The MOVE-JIA Trial
Brief Title: Optimizing Treatment for Patients With Juvenile Idiopathic Arthritis in Sustained Remission: The MOVE-JIA Trial
Acronym: MOVE-JIA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other); South-Eastern Norway Regional Health Authority (Other); Remedy (Industry)
Responsible Party: Principal Investigator, Anna-Birgitte Aga, Coordinating Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-513017-12-00; 2024-513017-12-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-17; First posted 2024-10-22 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-10

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: JIA; maintenance treatment; medication withdrawal; withdrawal
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Methotrexate; Tumor Necrosis Factor Inhibitors

STUDY DESIGN:
Intervention Model Description: Researcher initiated, randomized controlled, 3-arm, parallel group, national, multicenter clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stable treatment (Active Comparator): Stable treatment with methotrexate and TNFi
  Interventions: Drug: Methotrexate; Drug: TNF Inhibitor
- Methotrexate withdrawal (Experimental): Gradual withdrawal of methotrexate
  Interventions: Drug: Methotrexate
- TNFi withdrawal (Experimental): Gradual withdrawal of TNFi
  Interventions: Drug: TNF Inhibitor

INTERVENTIONS:
Drug: Methotrexate — Gradual withdrawal of the medication
  Arms: Methotrexate withdrawal; Stable treatment
Drug: TNF Inhibitor — Gradual withdrawal of the medication
  Arms: Stable treatment; TNFi withdrawal

SUMMARY:
The goal of this clinical trial is to compare three different maintenance and step-down treatment strategies in children and adolescents with juvenile idiopathic arthritis in sustained remission. The main questions it aims to answer are:

* Is the proportion of study participants with a disease flare different between each of the two drug withdrawal arms and the stable treatment arm during 12 months?
* Does the proportion of study participants with a disease flare differ between the two drug withdrawal arms during 12 months?
* How long time does it take before a disease flare occurs, and how long does it take before disease remission is reestablished for participants in the different treatment arms?

Participants will be randomized to either A) continued stable treatment with methotrexate and tumor-necrosis alpha inhibitor (TNFi); B) gradual withdrawal of methotrexate while continued stable dose TNFi; or C) gradual withdrawal of TNFi.

Participants will be examined every 4 month, and with extra visits if they experience increased symptoms or suspect a disease flare. If a flare occurs, the medications received at study inclusion will be restarted.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 2-<18 years of age at the time of signing the informed consent.
2. Fulfilment of the International League of Associations for Rheumatology (ILAR) classification criteria for non-systemic Juvenile Idiopathic Arthritis (JIA).
3. Inactive disease for ≥12 months documented at a minimum of 2 consecutive visits and documented inactive disease according to Wallace criteria at inclusion, and no active uveitis for ≥24 months.
4. Stable treatment with methotrexate and Tumor Necrosis Factor inhibitor (TNFi) for ≥6 months. Weight adjustments permitted.
5. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).
6. Male participants: No contraceptive measures necessary.
7. Female participants: contraception guidance for women of childbearing potential (WOCP).

Exclusion Criteria:

1. Chronic widespread pain syndrome
2. Major comorbidity including uncontrolled infectious, neurological or mental disease, malignant disease, severe heart failure, severe renal failure, active ulcus ventriculi, and uncontrolled diabetes mellitus.
3. Use of oral, intra-articular, intramuscular or intravenous corticosteroids due to JIA less than 12 months prior to randomization.
4. Participating in an ongoing clinical randomized study..
5. Drug/alcohol abuse which hampers adherence to the study protocol as based on the investigators judgement.
6. Language barriers that hamper adherence to the study protocol.
7. Pregnancy or breastfeeding.
8. Any condition that in the view of the investigator would suggest that the patient is unable to comply with the study protocol and procedures.
9. Unwillingness to use safe contraception for sexually active WOCP.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with disease flare | 4, 8 and 12 months
  Disease flare is defined as a combination of: A clinical significant increase in Juvenile Arthritis Disease Activity Score 27 (JADAS-27*) ≥1.7 from baseline AND active joints ≥1 (swollen, or tender + limited range of motion) OR consensus between treating physician and participant/parents that a clinically significant flare has occurred with need of intensification of antirheumatic treatment.
  *JADAS-27 is a composite measure of juvenile idiopathic arthritis (JIA) disease activity, calculated as a sum of scores from four components giving a score of 0-57. The components included are physician global assessment of disease activity, parent/patient's global assessment of well-being, active joint count of 27 joints and erythrocyte sedimentation rate (ESR) normalized to a 0-10 scale.
Proportion of patients with disease flare between two different withdrawal strategies | 4, 8 and 12 months
  Disease flare is defined as a combination of: A clinical significant increase in Juvenile Arthritis Disease Activity Score 27 (JADAS-27*) ≥1.7 from baseline AND active joints ≥1 (swollen, or tender + limited range of motion) OR consensus between treating physician and participant/parents that a clinically significant flare has occurred with need of intensification of antirheumatic (DMARD) treatment.
  *JADAS-27 is a composite measure of JIA disease activity, calculated as a sum of scores from four components giving a score of 0-57. The components included are physician global assessment of disease activity, parent/patient's global assessment of well-being, active joint count of 27 joints and ESR normalized to a 0-10 scale.

SECONDARY OUTCOMES:
Time to disease flare | 4, 8 and 12 months
  JADAS-27, physician's global assessment of diseasae activity, paren't/patient's global assessment, swollen, tender and range of motion joint count (assessed in 71 joints), ESR/CRP, consensus between treating physiciand and patient/parents (uveitis, arthritis on imaging, psoriasis, inflammatory back pain, enthesitis, other; yes/no)
  *JADAS-27 is a composite measure of JIA disease activity, calculated as a sum of scores from four components giving a score of 0-57. The components inculded are physician global assessment of disease activity, parent/patient's global assessment of well-being, active joint count of 27 joints and ESR normalized to a 0-10 scale.
Time to regain inactive disease by the Wallace definition* after flare | 4, 8 and 12 months
  JADAS-27, Wallace inactive disease*, physician's global assessment of disease activity, paren't/patient's global assessment, swollen, tender and range of motion joint count (assessed in 71 joints), ESR/CRP, consensus between treating physiciand and patient/parents (uveitis, arthritis on imaging, psoriasis, inflammatory back pain, enthesitis, other; yes/no).
  *Wallace inactive disease: No active arthritis, no active uveitis, no morning stiffness >15 minutes, no systemic features (fever/rash/serositis/splenomegaly/lymphadenopathy due to JIA), a physician global assessment of disease activity 0 on a 0-100 scale) and normalization of C-reactive protien (CRP) and ESR.
Physician global assessment of disease activity | 4, 8 and 12 months
  Physician global assessment of disease activity is measured on a 100 mm visual analogue scale (VAS). The anchors of the scale are "very well" to "very poor".
Disease activity assessed by joint count | 4, 8 and 12 months
  In total 68 joints will be evaluated for swelling, 75 joints/joint areas will be evaluated for tenderness and 70 joints/joint areas will be examined for limitation of motion. JADAS10, JADAS27 and JADAS71 and 71-joint count will be computed from this examination
Patient's/parent's global assessment of well-being | 4, 8 and 12 months
  Patient's/parent's global assessment of well-being will be assessed on a 100 mm visual analouge scale.
Concentration of Erythrocyte sedimentation rate (ESR), | 4, 8 and 12 months
  Erythrocyte sedimentation rate (ESR), will be measured at all clinical visits
Concentration of C-reactive protein (CRP) | 4, 8 and 12 months
  C-reactive protein (CRP) will be measured at all clinical visits
Numbers and type of adverse events (AE) | 4, 8 and 12 months
  Assessment of AE, serious AE and suspected unexpected serious adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Birgitte Aga, MD PhD, Principal Investigator — Oslo University Hospital
Locations (7):
- Norway (7):
  - Haukeland University Hospital, Bergen
  - Drammen Hospital, Drammen
  - Hospital of Southern Norway Hospital Trust, Kristiansand
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital of North Norway, Tromsø
  - St. Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
A de-identified patient data set can be made available to researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 10 years
Access Criteria: The data will only be made available after submission of a project plan outlining a reasonable request and any proposed analyses, and will have to be approved by the the MOVE-JIA steering group. Project proposals can be submitted to the corresponding author. Data sharing will have to follow appropriate regulations.